CLINICAL TRIAL: NCT02413580
Title: A Multicenter, Prospective, Open-label, Non-controlled Clinical Trial to Assess the Efficacy and Safety of Immune Globulin (Human), 10% Caprylate/Chromatography Purified (IGIV-C) in Patients With Myasthenia Gravis Exacerbations
Brief Title: A Study to Assess the Efficacy and Safety of IGIV-C in Patients With Myasthenia Gravis Exacerbations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTI1305
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Myasthenia Gravis Exacerbations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IGIV-C Treatment (Experimental): In this arm, subjects with myasthenia gravis exacerbations were treated with an IV dose of 2 g/kg of IGIV-C, which was administered over 2 consecutive days at a dose of 1 g/kg per day.
  Interventions: Biological: IGIV-C

INTERVENTIONS:
Biological: IGIV-C — An IV dose of 2 g/kg of IGIV-C was administered over 2 consecutive days at a dose of 1 g/kg per day.

SUMMARY:
This was a multicenter, prospective, open-label, non-controlled study to assess the efficacy and safety of an IV dose of 2 g/kg of IGIV-C in subjects with MG exacerbations.

DETAILED DESCRIPTION:
The study consisted of a single dose course of IGIV-C treatment followed by 28-days of post-infusion assessments. The total duration of study participation for each subject was up to 28 ± 2 days. Approximately 50 subjects, ages 18 or greater, were planned to be enrolled in the study and receive a single, total dose of 2 g/kg of IGIV-C over 2 consecutive days (dose of 1 g/kg per day) across multiple centers in Argentina, Canada, Europe, and South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Was male or female aged ≥18 years.
* Subjects must be willing and able to provide written informed consent (if applicable, a legally authorized representative may provide informed consent on behalf of the subject).
* Subjects who met the clinical criteria for diagnosis of MG with an exacerbation defined as worsening of MG symptoms as defined by an Myasthenia Gravis Foundation of America (MGFA) classification IVb or V.
* Subjects on long-term (8 weeks) corticosteroid treatment for MG.
* Female subjects of child-bearing potential must have a negative test for pregnancy (human chorionic gonadotropin [HCG]-based assay).
* Subjects must be willing to comply with all aspects of the clinical trial protocol, including blood sampling and long-term storage of extra samples, for the entire duration of the study.

Exclusion Criteria:

* Subjects who had received immune globulin treatment given by IV, subcutaneous or intramuscular route within the last 30 days.
* Subjects with documentation of a lack of clinical response to intravenous immunoglobulin (IVIg) therapy for MG.
* Subjects documented positive for antibodies directed against Muscle specific kinase (MuSK).
* Subjects with corticosteroid (CS) treatment initiated within the last 8 weeks or modified within the last 2 weeks.
* Subjects with plasma exchange (PLEX) within the last 30 days.
* Subjects with MG exacerbation attributable to change in medication or infection or evident infection as defined by, but not limited to, the presence of at least one of the following diagnostic features: 1) axillary temperature ≥38°C, 2) positive blood culture of infective microorganism, 3) white blood cell count >12×10^9/L and differential white blood cell count of >10% band neutrophils (>1.2×10^9/L), and 4) pulmonary infiltrate with consolidation on chest X-ray. Alternatively, other signs and symptoms may be considered for the diagnosis of evident infection according to the Investigator's judgement.
* Subjects with inadequate venous access.
* Subjects with a history of anaphylactic reactions or severe reactions to any blood-derived product.
* Subjects with a history of intolerance to any component of the investigational products.
* Subjects with a documented diagnosis of thrombotic complications to polyclonal IVIG therapy in the past.
* Subjects with a history of recent (within the last year) myocardial infarction, stroke or uncontrolled hypertension.
* Subjects who suffered from uncontrolled congestive heart failure, embolism or documented electrocardiogram (ECG) changes indicative of myocardial ischemia or atrial fibrillation.
* Subjects with current known hyperviscosity or hypercoagulable state.
* Subjects currently receiving anti-coagulation therapy.
* Subjects with a history of chronic alcoholism or illicit drug abuse (addiction) in the 12 months preceding the Baseline Visit.
* Subjects currently receiving, or having received within 3 months prior to the Baseline Visit, any investigational medicinal product or device.
* Subjects with a known Immunoglobulin A (IgA) deficiency and anti-IgA serum antibodies.
* Subjects with renal impairment (i.e., serum creatinine exceeds more than 1.5 times the upper limit of normal [ULN] for the expected normal range for the testing laboratory).
* Subjects with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels exceeding more than 2.5 times the ULN for the expected normal range for the testing laboratory.
* Subjects with haemoglobin levels <9 g/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-03; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- Argentina (3):
  - Hospital Italiano, Buenos Aires
  - Hospital General de Agudos Dr. J. M., Buenos Aires
  - Hospital Cordoba, Córdoba
- Belgium (2):
  - AZ St Lucas Gent, Ghent, East Flanders
  - UZ Leuven, Leuven
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - University Health Network (UHN) - Toronto General Hospital, Toronto, Ontario
- Czechia (3):
  - Fakultni nemocnice Brno, Neurologicka klinika, Brno
  - Fakultni nemocnice Ostrava, Neurologická klinika, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
- East Tallinn Central Hospital, Tallinn, Estonia
- France (6):
  - Hopital Neurologique Pierre Wertheimer, Bron, Lyon
  - Hôpital Albert Michallon, Grenoble
  - Hopital Roger Salengro, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Hautepierre Strasbourg, Strasbourg
  - CHU de Toulouse - Hôpital Purpan, Toulouse
- Hungary (5):
  - Jahn Ferenc Del-Pesti Korhaz, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Nyíregyháza
  - University of Szeged, Faculty of Medicine, Szeged
  - Zala Megyei Korhaz, Zalaegerszeg
- Riga East Clinical University Hospital, Riga, Latvia
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- Romania (2):
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu-Mures, Târgu Mureş
- Russia (3):
  - State Budgetary Institution of Healthcare of Nizhniy Novgorod region. Nizhniy Novgorod Regional Clinical Hospital named after N.A.Semashko, Nizhny Novgorod
  - Saint-Petersburg State Budgetary Institution of Healthcare. City Multi-field Hospital # 2, Saint Petersburg
  - State Budgetary Institution of Healthcare "Samara Regional Clinical Hospital. V.D.Seredavin, Samara
- Groote Schuur Hospital,, Cape Town, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- IGIV-C Treatment: An IV dose of 2 g/kg of IGIV-C was administered in subjects with myasthenia gravis exacerbations.
  IGIV-C: an IV dose of 2 g/kg of IGIV-C was administered as 2 doses of 1 g/kg on two consecutive days
Period: Overall Study
Arm/Group | IGIV-C Treatment
Started | 49
Completed | 46
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: The demographic data are from the Safety population that consisted of all 49 subjects who were infused with any amount of study drug.
Arm/Group | IGIV-C Treatment
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 40
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: year] | 47.3 (15.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 44
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3
  Argentina | 3
  Latvia | 10
  Romania | 5
  Belgium | 6
  Czechia | 4
  Poland | 4
  South Africa | 2
  France | 2
  Russia | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Quantitative Myasthenia Gravis (QMG) Scale Score
Description: Mean Change in Quantitative Myasthenia Gravis (QMG) Scale Score from Baseline (Day 0) to Day 14. The minimum and maximum scores of the QMG Scale are 0 and 39, respectively, and a higher score means a worse outcome.
Time Frame: From Baseline (Day 0) to Day 14
Population: The primary efficacy analysis of change in the score of MG symptoms as measured by the change in QMG score from Baseline (Day 0) to Day 14 in the Evaluable population which consisted of all subjects who received the entire dose of Investigational Product (2 g/kg over 2 consecutive days) and had valid baseline and Day 14 QMG Score measurements.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IGIV-C Treatment
Number analyzed (Participants) | 43
score on a scale | -6.4 (5.15)
Statistical Analysis 1: Comparison: IGIV-C Treatment; Test type: Other — The hypothesis test is to test the null hypothesis: H0: μd = 0 versus alternative hypothesis Ha: μd ≠ 0 where μd is the mean change from Baseline to Day 14. The Shapiro-Wilk test is used to test the normality. If the assumptions for parametric test are met, a paired t-test (comparison between the pre- and post-treatment) is used to test for the treatment effect. Otherwise, a non-parametric test (Wilcoxon signed rank test) is used; p < 0.001, Paired t-test; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-7.957 to -4.787]

2. Secondary Outcome: Percentage of Subjects With Clinical Improvement Assessed by QMG
Description: The percentage of subjects with clinical improvement at Day 14 as assessed by the Quantitative Myasthenia Gravis (QMG) scale in the Evaluable population is presented, in which clinical improvement is defined as at least 3-point decrease in QMG score from Baseline (Day 0) to Day 14. The minimum and maximum scores of the QMG scale are 0 and 39, respectively, and a higher score means a worse outcome.
Time Frame: Baseline (Day 0) to Day 14
Population: The percentage of subjects with clinical improvement at Day 14 as assessed by the QMG scale in the Evaluable population is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | IGIV-C Treatment
Number analyzed (Participants) | 43
Participants | 33

3. Secondary Outcome: Percentage of Subjects With Clinical Improvement Assessed by MG-Activities of Daily Living (MG-ADL) Scale
Description: The percentage of subjects with clinical improvement at Day 14 as assessed by the MG-ADL Scale in the Evaluable population is presented, in which clinical improvement is defined as at least 2-point decrease in the MG-ADL score. The minimum and maximum scores of the MG-DAL scale are 0 and 24, respectively, and a higher score means a worse outcome.
Time Frame: Baseline (Day 0) to Day 14
Population: The percentage of subjects with clinical improvement at Day 14 as assessed by the MG-ADL in the Evaluable population is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | IGIV-C Treatment
Number analyzed (Participants) | 43
Participants | 38

4. Secondary Outcome: Percentage of Subjects With Clinical Improvement Assessed by the MG Composite
Description: The percentage of subjects with clinical improvement at Day 14 as assessed by the MG Composite scale in the Evaluable population is presented in which clinical improvement is defined as at least 3-point decrease in the MG Composite score. The minimum and maximum scores of the MG Composite scale are 0 and 50, respectively, with a higher score meaning a worse outcome.
Time Frame: Baseline (Day 0) to Day 14
Population: The percentage of subjects with clinical improvement at Day 14 as assessed by the MG Composite scale in the Evaluable population is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | IGIV-C Treatment
Number analyzed (Participants) | 43
Participants | 37

ADVERSE EVENTS:
Time Frame: Subjects with MG exacerbations not attributable to an infection or change in medication were planned to receive 2 g/kg of IGIV-C on Day 0 (Baseline) and on Day 1 (dosed as 1 g/kg per day), followed by 28 days of post-infusion assessments. During this 30-day period, the adverse event data were collected.
Arm/Group | IGIV-C Treatment
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 30/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C Treatment (N=49)
Headache (Nervous system disorders) | 19 (21)
Influenza like illness (General disorders) | 3 (3)
Pyrexia (General disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT02413580/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT02413580/SAP_001.pdf